CLINICAL TRIAL: NCT03623568
Title: Pan-genotypic Direct Acting Antiviral Therapy in Donor HCV-positive to Recipient HCV-negative Kidney Transplant
Brief Title: Direct Acting Antiviral Therapy in Donor HCV-positive to Recipient HCV-negative Kidney Transplant
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: did not move forward with IRB approval, competing study
Sponsor: Raymond T. Chung, MD (Other)
Responsible Party: Sponsor-Investigator, Raymond T. Chung, MD, Director of Hepatology, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2018P001077
Record Dates: First submitted 2018-08-02; First posted 2018-08-09 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-05

CONDITIONS: Kidney Failure; Kidney Diseases; Hepatitis C
Keywords: CKD; HCV; Hepatitis C; Transplant
MeSH Terms: conditions — Renal Insufficiency; Kidney Diseases; Hepatitis C | interventions — glecaprevir; pibrentasvir; glecaprevir and pibrentasvir

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment with Mavyret (glecaprevir/pibrentasvir) for HCV (Experimental): 12 weeks of treatment with Mavyret
  Interventions: Drug: glecaprevir/pibrentasvir tablets

INTERVENTIONS:
Drug: glecaprevir/pibrentasvir tablets — 12 weeks of treatment with Mavyret
  Other Names: Mavyret

SUMMARY:
This is a proof of concept, single center study for the donation of HCV-positive kidney to HCV negative recipient patients, with preemptive, interventional treatment with 12 weeks of commercially available DAA therapy to prevent HCV transmission upon transplantation.

DETAILED DESCRIPTION:
The goal of this study is to determine if preoperative dosing and sustained administration of pan-genotypic DAA therapy after kidney transplantation prevents the transmission of hepatitis C virus (HCV) infection from an HCV positive donor kidney to an HCV naïve recipient.

ELIGIBILITY:
Inclusion Criteria:

* Met MGH transplant center criteria and already listed for kidney transplant
* No available living kidney donor
* Has ≤ 730 days (two years) of accrued transplant waiting time if blood type A and ≤ 1095 days of accrued transplant waiting time if blood type B or O.
* On chronic hemodialysis or peritoneal dialysis or has a glomerular filtration rate <15mL/min/1.73m2 at the time of screening
* Must agree to birth control. Women must agree to use birth control in accordance with Mycophenolate Risk Evaluation and Mitigation Strategy and at least one barrier method
* Weigh at least 50kg
* Serum ALT within normal limits with no history of liver disease
* Able to sign informed consent

Exclusion Criteria:

* AB blood type
* BMI > 35
* Any liver disease in recipient
* Pregnant or nursing (lactating) women
* Known allergy or intolerance to tacrolimus that would require administration of cyclosporine rather than tacrolimus given the known drug-drug interaction between cyclosporine and Mavyret
* Cardiomyopathy (LV ejection fraction < 50%)
* Albumin < 3g/dl or platelet count < 75 x 103/mL
* Positive donor specific antibodies or positive cross match deemed to be clinically relevant and increasing risk of rejection per the transplant surgeon or nephrologist
* Positive donor specific antibodies or positive cross match deemed to be clinically relevant and increasing risk of rejection per the transplant surgeon or nephrologist
* HCV RNA positive
* Hepatitis B surface antigen positive
* Any known liver disease or elevated liver transaminases
* Patients with primary focal segmental glomerulosclerosis (FSGS), FSGS recurring after previous transplant, or disease process with increased risk of causing early graft failure as assessed by the transplant nephrologist and/or the investigator team
* Any contra-indication to kidney transplantation per MGH center protocol
* Patients on the following medications who cannot stop therapy: carbamazepine, rifampin, St. John's wort, and ethinyl estradiol-containing oral contraceptives.

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-02-15 (Estimated); Primary Completion 2020-12-31 (Estimated); Study Completion 2021-04-15 (Estimated)

PRIMARY OUTCOMES:
Undetectable HCV RNA in blood | 12 weeks post treatment
  Negative HCV viral RNA at 12 weeks after the last dose of treatment as determined by blood test

SECONDARY OUTCOMES:
Safety (based on number of adverse events and out of range lab values) of DAA therapy in patients undergoing kidney transplantation) | 12 weeks post treatment
  Safety of Mavyret therapy in the kidney transplant patient will be monitored by quantifying the number of treatment related adverse events per patient and evaluating out of range laboratory results as compared to baseline/pretreatment values per patient.
Tolerability (based on number of adverse events and out of range lab values) of DAA therapy in patients undergoing kidney transplantation | 12 Weeks post treatment
  Tolerability of Mavyret therapy in the kidney transplant patient will be monitored by quantifying the number of treatment related adverse events per patient and evaluating out of range laboratory results as compared to baseline/pretreatment values per patient.

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
Anticipate to share coded data with collaborators
Supporting Information: Study Protocol
Time Frame: Anticipate data would be available to share within 6 months after the final patient completes the study.
Access Criteria: Coded data would be shared with collaborators who have received IRB approval to use the data and have been approved by the PI for their collaboration.